CLINICAL TRIAL: NCT04713332
Title: Effectiveness of Vitamin E and Molecular Hydrogen-Rich Water on Radiation Therapy-Induced Adverse In Adult Patients With Rectal Carcinoma in Al-Quds, Palestine
Brief Title: Effectiveness of Vitamin E and Hydrogen-Rich Water on Radiation Therapy-Induced Adverse In Patients With Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jordan (Other)
Collaborators: Slovak Academy of Sciences (Other Government); Al-Quds University (Other)
Responsible Party: Principal Investigator, Ziad Abuawad, PhD Candidates in Human Nutrition and Dietetics, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCT-2021
Record Dates: First submitted 2021-01-13; First posted 2021-01-19 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Radiation-induced Injuries in Patients With Rectal Cancer
MeSH Terms: interventions — Vitamin E; alpha-Tocopherol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- vitamin E (Active Comparator): Oral intake of Vitamin E treatment will be given on a daily basis in a single-blind manner one day before the first day of RT and continued for 8 weeks. Patients in the group receiving 500 IU of d-alpha-tocopherol capsules orally (3 times daily).
  Interventions: Dietary Supplement: Vitamin E
- Hydrogen rich water (Active Comparator): Oral intake of HRW (2 ppm) treatment will be given on a daily basis in a single-blind manner one day before the first day of RT and continued for 8 weeks. The group of patients receiving Hydrogen water took an amount of 250 ml orally 3 times a day.
  Interventions: Dietary Supplement: Hydrogen rich water
- placebo (Placebo Comparator): Oral intake of placebo will be given on a daily basis in a single-blind manner one day before the first day of RT and continued for 8 weeks. The placebo group received 3 soft gel placebo capsules containing gelatin three times a day.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Vitamin E — Members of the vitamin E family are hydrophobic fat-soluble compounds found in a variety of food sources such as vegetable oils, fruits, and vegetables consumed through diet. Vitamin E exists in 8 isoforms, a, b, g, d-tocopherol, and a, b, g, d-tocotrienol. The recommended daily allowance for adults is 15 mg per day for alpha-tocopherol, an amount which is easily met by dietary sources, and 30 mg per day for synthetic all-rac-alpha-tocopherol. The upper limit for intake is 1,000 mg per day. Very often, the dosage of vitamin E is given in international units (IU) as capsules, with a typical dose being 400 IU per day, which is above the recommended daily allowance. The health benefits of consuming vitamin E through diet or supplementation are believed to be for its antioxidant properties as a peroxyl radical scavenger. Vitamin E protects cells from cell damage caused by free radicals that damage cell membranes through lipid oxidation leading to DNA damage and cancer development.
  Other Names: 500 IU of d-alpha-tocopherol
  Arms: vitamin E
Dietary Supplement: Hydrogen rich water — Molecular hydrogen is a new medical gas that can be dissolved in water and administered through drinking, inhalation, baths, intravenous drip. A growing body of evidence indicates that hydrogen, as a novel antioxidant, scavenges hydroxyl radical and peroxynitrite. In contrast to other antioxidants, gaseous molecular hydrogen efficiently penetrates cytoplasmic membranes and targets intracellular organelles, largely owing to its small size and neutral electricity. Thus, hydrogen has been suggested as a suitable candidate for the therapeutic strategies for various diseases, including certain types of cancer. Hydrogen has emerged as a promising cancer remedy as a preventative agent or in combined therapy with anticancer drugs. Hydrogen water consumption might mitigate the side effects of anticancer drugs by decreasing oxidative stress and ameliorating metamorphosis due to decreased apoptosis.
  Arms: Hydrogen rich water
Dietary Supplement: placebo — Placebo containing gelatin is made by cooking down the protein collagen found in the skin, hooves, connective tissues, and bones of animals. The cooking process breaks down the bonds between proteins to make smaller, more bioavailable building blocks that your body can easily absorb. Like collagen, gelatin is packed with beneficial amino acids, especially the anti-aging superstar's glycine and proline, which are lacking in the standard Western diet. These amino acids make gelatin especially powerful for healing skin, gut, and joint damage. Because collagen and gelatin come from the same source, they have identical amino acid profiles
  Arms: placebo

SUMMARY:
Controlled studies investigating the effects of vitamin E or H2 water or comparing their effectiveness on radiation therapy-induced injuries in RC patients are generally lacking. The present study hypothesis the following: (1) Pre - radiation therapy administration of vitamin E to patients with rectal carcinoma will provide radioprotection for exposed healthy tissues. (2) Consumption of H2 water by patients with rectal carcinoma undergoing RT will reduce the side effects of this modality. (3) Rectal cancer patients receiving H2 water will show better biological improvement than those receiving only vitamin E, i.e., H2 water is more effective antioxidant than vitamin E. (4) The proposed radiation countermeasures will not compromise the anti-tumor effects.

ELIGIBILITY:
Inclusion Criteria:

* - Men or women.
* Older than 18 years.
* Histologically proven adenocarcinoma of the rectum.
* Underwent radiotherapy.
* Absence of any psychological, and sociological condition that potentially affects the compliance with the study protocol and follow-up schedule.

Exclusion Criteria:

* The use of anticoagulant and antiplatelet agents.
* Any disease of disorder capable of contraindicating the absorption of Vitamin E or Hydrogen water in the body of a patient being investigated.
* No known history of problems absorbing fats (e.g., Crohn disease, cystic fibrosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-06 (Actual); Primary Completion 2021-03-08 (Estimated); Study Completion 2021-05-08 (Estimated)

PRIMARY OUTCOMES:
total blood count | One day before the first day of radiation exposure (initial data) and 2, 6 and 8 weeks post radiation exposure
  A hematology analyzer is commonly used to investigate changes in hematological parameters, which vary in response to systemic changes. These hematological parameters include WBCs, which defend the body against foreign invaders; their numbers increase during inflammation. RBCs contain hemoglobin, which carries oxygen to the tissues. Platelets have a hemostatic function. During injury, they gather at the site of damage in blood vessels and form a primary platelet plug. Bleeding occurs when the platelet count decreases.
Nuclear factor erythroid 2-related factor 2 (Nrf2) | One day before the first day of radiation exposure (initial data) and 2, 6 and 8 weeks post radiation exposure
  Nrf2, a basic leucine-zipper containing transcription factor that plays a key role in the regulation of the production and expression of antioxidant genes in the body. Nrf2 usually combines with the ARE, which is the upstream promoter region of SOD, CAT, GPx, etc. After combination, the enzyme complex upregulate the expression of a serious endogenous protective antioxidant genes in the tissue, thereby maintaining the balance of oxidation and antioxidant levels of the cells.
Superoxide dismutases (SOD) | One day before the first day of radiation exposure (initial data) and 2, 6 and 8 weeks post radiation exposure
  SODs are a group of metalloenzymes that are found in all kingdoms of life. SODs form the front line of defense against reactive oxygen species (ROS)-mediated injury. These proteins catalyze the dismutation of superoxide anion free radical (O2-) into molecular oxygen and hydrogen peroxide (H2O2) and decrease O2- level which damages the cells at excessive concentration. This reaction is accompanied by alternate oxidation-reduction of metal ions present in the active site of SODs. During oxidative damage, the level of this enzyme within the tissues is elevated in order to protect them. SOD converts O2- into H2O2.
Catalase (CAT) | One day before the first day of radiation exposure (initial data) and 2, 6 and 8 weeks post radiation exposure
  CAT is a common enzyme found in nearly all living organisms, which are exposed to oxygen. The first function assigned to catalase is the transformation of hydrogen peroxide into oxygen and water. It thus plays an important role in defending cells against oxidative damage by degrading hydrogen peroxide. Catalase can modulate the growth rate by various mechanisms, the first obviously being its ability to detoxify H2O2. The second is its ability to bind and protect certain proteins from potential oxidative damage, which in turn are involved in the processes of proliferation and migration. As shown by many reports, catalase and mitochondrial superoxide dismutase control cell growth and migration processes in cancer cells.
Glutathione S-transferase (GST) | One day before the first day of radiation exposure (initial data) and 2, 6 and 8 weeks post radiation exposure
  GST isoenzyme superfamilies detoxify a wide-range of toxic chemicals and environmental substances are extensively expressed in mammalian tissues. GSTs play a key role in the deactivation of reactive oxygen species (ROS) and the metabolism of lipids, chemotherapeutic agents. GSTs are mainly involved in conjugation of reduced glutathione (GSH) with diverse substrates specificity and it is possible that genetic variations in these enzymes will influence cellular response to the environmental agents. GSTs are overexpressed in response to a chemical or oxidative stress as an adaptive physiology and upregulated in cancerous state of organ or tissue. GSTs are essentially involved in susceptibility to various forms of cancer as they are vital in detoxification mechanism to metabolize the environmental carcinogens.
Malondialdehyde (MDA) | One day before the first day of radiation exposure (initial data) and 2, 6 and 8 weeks post radiation exposure
  MDA is one of the consequences of uncontrolled oxidative stress is cells, tissues, and organs injury caused by oxidative damage. It has long been recognized that high levels of free radicals or reactive oxygen species (ROS) can inflict direct damage to lipids. MDA is an end-product generated by decomposition of arachidonic acid and larger PUFAs, through enzymatic or nonenzymatic processes. MDA is highly reactive, capable of inhibiting enzymes that protect cells against the harmful effects of oxidative stress.
Tumor necrosis factors (TNF) | One day before the first day of radiation exposure (initial data) and 2, 6 and 8 weeks post radiation exposure
  TNF refer to a group of cytokines which are mainly secreted by monocytes/macrophages. While it was first recognized for its anti-tumor activity, TNF has since been identified as a highly pleiotropic cytokine that mediates multiple cellular processes including inflammation, cell differentiation, cell survival and proliferation, and apoptosis. The master pro-inflammatory cytokine, TNF, has been shown to modulate multiple signaling pathways, with wide-ranging downstream effects. TNF plays a vital role in the typical immune response through the regulation of a number of pathways encompassing an immediate inflammatory reaction with significant innate immune involvement as well as cellular activation with subsequent proliferation and programmed cell death or necrosis.
Matrix metalloproteinases(MMPs) | One day before the first day of radiation exposure (initial data) and 2, 6 and 8 weeks post radiation exposure
  MMPs are members of metzinc in group of zinc dependent endopeptidases which are responsible for degrading and remodeling of extracellular matrix (ECM) during organogenesis, wound healing, angiogenesis, apoptosis, cell proliferation and cancer progression. The expression and activity of MMPs in adult tissues is normally quite low, but increases significantly in various pathological conditions that may lead into unwanted tissue destruction, such as inflammatory diseases, tumour growth and metastasis. MMPs are produced by multiple tissues and cells. MMPs are secreted by connective tissue, pro-inflammatory, and uteroplacental cells.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Numan, Professor, Study Chair — The University of Jordan; Jan Slezak, Professor, Study Chair — The Slovak Academy of Sciences
Locations (1):
- Augusta Victoria Hospital, East Jerusalem, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No